CLINICAL TRIAL: NCT03988088
Title: A Phase 1, Open-Label, Single-Dose Pharmacokinetic Study of Lasmiditan in Pediatric Patients With Migraine
Brief Title: A Study of Lasmiditan (LY573144) in Children Aged 6 to 17 With Migraine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16932; H8H-MC-LAHX (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-05-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lasmiditan (Experimental): Participants with lower body weight (15 to ≤40 kilograms (kg)) received single oral dose of 100 milligrams (mg) Lasmiditan in Cohort 1 and higher body weight (>40 to ≤55 kg) participants received single oral dose of 200 mg Lasmiditan in Cohort 2.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally.
  Other Names: LY573144

SUMMARY:
The purpose of the study is the measure the levels of lasmiditan in the body of children aged 6 to 17 with migraine. The study also will also examine the safety and tolerability of lasmiditan in children aged 6 to 17 with migraine.

The study will last about 6 weeks, and includes 4 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a history of migraine headaches for more than 6 months
* Participants must have a history of 2 to 15 migraine headaches per month in the past 2 months
* Participants must weigh between 15 and 55 kilograms (kg)
* Participants must not have a migraine headache on the day of lasmiditan administration

Exclusion Criteria:

* Participants must not be pregnant or nursing
* Participants must not have any acute, serious, or unstable medical condition

  * Participants must not be actively suicidal or at significant risk for suicide, in the opinion of the investigator
* Participants must not be on a medicine that acts in the brain and spinal cord

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-01-19 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (8):
  - Perserverance Research Center, Scottsdale, Arizona
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Meridien Research, Bradenton, Florida
  - Meridien Research, Maitland, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Japan (2):
  - Kurume Clinical Pharmacology Clinic, Kurume, Fukuoka
  - Clinical Research Hospital, Tokyo, Shinjuku-Ku, Tokyo
- San Jorge Children and Women's Hospital- Shipping Location, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tsai M, Nery ESM, Kerr L, Khanna R, Komori M, Dennehy EB, Wilbraham D, Winner P. Pharmacokinetics, Safety, and Tolerability of Lasmiditan in Pediatric Patients with Migraine. Clin Pharmacokinet. 2021 Jun;60(6):819-828. doi: 10.1007/s40262-020-00966-z. Epub 2021 Feb 10. PMID 33565026
- See also: A Study of Lasmiditan (LY573144) in Children Aged 6 to 17 With Migraine — https://www.lillytrialguide.com/en-US/studies/migraine/LAHX#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 3-month open-label extension addendum was to evaluate safety and tolerability.
Groups:
- 100 Milligrams (mg) Lasmiditan: Participants with lower body weight (15 to ≤40 kilograms (kg)) received single oral dose of 100 mg Lasmiditan.
- 200 mg Lasmiditan: Participants with higher body weight (>40 to ≤55 kg) received single oral dose of 200 mg Lasmiditan.
- 50 mg Lasmiditan-Addendum: Participants with lower body weight (15 to ≤40 kg) received single oral dose of 50 mg Lasmiditan.
- 100 mg Lasmiditan-Addendum: Participants with higher body weight (>40 to ≤55 kg) received single oral dose of 100 mg Lasmiditan.
Period: Single-Dose Pharmacokinetic Study
Arm/Group | 100 Milligrams (mg) Lasmiditan | 200 mg Lasmiditan | 50 mg Lasmiditan-Addendum | 100 mg Lasmiditan-Addendum
Started | 11 | 7 | 0 | 0
Completed | 11 | 6 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Open-Label Addendum
Arm/Group | 100 Milligrams (mg) Lasmiditan | 200 mg Lasmiditan | 50 mg Lasmiditan-Addendum | 100 mg Lasmiditan-Addendum
Started | 0 | 0 | 2 (The US participants had the option to enter this optional 3-month open-label extension addendum.) | 2 (The US participants had the option to enter this optional 3-month open-label extension addendum.)
Completed | 0 | 0 | 1 | 2
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received study drug.
Groups:
- 100 mg Lasmiditan: Participants with lower body weight (15 to ≤40 kilograms (kg)) received single oral dose of 100 mg Lasmiditan.
- Total: Total of all reporting groups
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.09 (2.02) | 14.00 (2.65) | 11.00 (3.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 10
  Japan | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lasmiditan
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lasmiditan.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 8, 12 and 24 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 11 | 7
nanograms per milliliter (ng/mL) | 362 (46.7) | 426 (43.5)

2. Primary Outcome: PK: Area Under the Concentration-Versus-Time Curve (AUC) From Time Zero to Infinity (AUC[0-∞]) of Lasmiditan
Description: PK: Area Under the Concentration-Versus-Time Curve (AUC) from Time Zero to Infinity (AUC[0-∞]) of Lasmiditan.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 8, 12 and 24 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(ng*hr/mL)
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 11 | 6
nanograms*hours per milliliter(ng*hr/mL) | 2050 (38.4) | 2590 (13.7)

ADVERSE EVENTS:
Time Frame: Up To 3.5 Months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 100 mg Lasmiditan | 200 mg Lasmiditan | 50 mg Lasmiditan-Addendum | 100 mg Lasmiditan-Addendum
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 3/11 | 5/7 | 0/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mg Lasmiditan (N=11) | 200 mg Lasmiditan (N=7) | 50 mg Lasmiditan-Addendum (N=2) | 100 mg Lasmiditan-Addendum (N=2)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (2)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol: LAHX 05 Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT03988088/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03988088/SAP_001.pdf
  • Study Protocol: LAHX Protocol Addendum (1.1) (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT03988088/Prot_002.pdf